CLINICAL TRIAL: NCT05558176
Title: Intrapartum Sildenafil Citrate to Prevent Non Reassuring Foetal Status Among Parturients Delivering at LAUTECH Teaching Hospital, Ogbomoso, a Randomised Controlled Trial
Brief Title: Intrapartum Sildenafil Citrate to Prevent Non Reassuring Foetal Status Among Parturients Delivering at Term
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ladoke Akintola University of Technology Teaching Hospital, Ogbomoso (Other)
Responsible Party: Principal Investigator, Muritala Wakeel Okanlawon, Doctor, Lecturer/Consultant Obstetrician and Gynaecologist, Ladoke Akintola University of Technology Teaching Hospital, Ogbomoso
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LadokeAkintolaU
Record Dates: First submitted 2022-08-28; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Foetal Hypoxia
Keywords: foetal compromise; foetal distress; caesarean section
MeSH Terms: conditions — Fetal Hypoxia; Fetal Distress | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Selection of patients into each arm of the study will be through a computer generated sequence in a 1:1 ratio to receive either sildenafil citrate or placebo in variable blocks of up to six (Stata Statistical Software, Release 14; College Station, TX; StataCorp LP. StataCorp 2013) in a sealed opaque envelope. Each participant's study identification number will be recorded in the clinical notes.
  The packaging of the trial drugs will be carried out under sterile hygienic condition in the hospital pharmacy department by two of the hospital pharmacists who will be dedicated to the study, they will prepare sequentially ordered packs labelled with individual study identification numbers containing identical tablets of sildenafil citrate or placebo, they will be the only one who know which number is assigned to sildenafil citrate or placebo. The same brand of sildenafil citrate
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The packaging of the trial drugs will be carried out under sterile hygienic condition in the hospital pharmacy department by two of the hospital pharmacists who will be dedicated to the study, they will prepare sequentially ordered packs labelled with individual study identification numbers containing identical tablets of sildenafil citrate or placebo, they will be the only one who know which number is assigned to sildenafil citrate or placebo.
  Women, clinicians, and principal investigator will be unaware of allocation. Clinical staff managing the labour will be blinded to the ultrasound results and retained responsibility for all decisions regarding intrapartum care. At LTH Ogbomoso, all decisions for caesarean delivery are made by the obstetrics team under the supervision of consultant Obstetrician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil citrate arm (Active Comparator): The same brand of sildenafil citrate (VIAGRA, manufactured by Fareva Amboise Zone Industrielle, 29 route des Industries, 37530 Poce Sur Cisse, France, under authority of Pfizer Inc, NewYork, NAFDAC Reg NO: 04 - 1509, Batch No: 477209; Exp date: 11 - 2024) will be used in the course of the study.
  Women will receive the first dose of trial medication after transfer to the birth suite once diagnosed to be in labour with cervical dilatation < 8 cm. Sildenafil citrate will be given orally as a 50-mg dose 6 hourly to a maximum of 3 doses (150mg). Blood pressure will be monitored 15-30 minutes after each dose. Labour will be monitored with the aid of partograph, appropriate analgesic given in labour. Foetal heart rate monitoring will be performed in all cases by cardiotocograph or intermittent auscultation every fifteen minutes
  Interventions: Drug: Sildenafil citrate
- Placebo (Placebo Comparator): The placebo will be a vitamin C of the same size, colour and shape with sildenafil (Viagra).
  Interventions: Drug: Sildenafil citrate

INTERVENTIONS:
Drug: Sildenafil citrate — The same brand of sildenafil citrate (VIAGRA, manufactured by Fareva Amboise Zone Industrielle, 29 route des Industries, 37530 Poce Sur Cisse, France, under authority of Pfizer Inc, NewYork, NAFDAC Reg NO: 04 - 1509, Batch No: 477209; Exp date: 11 - 2024) will be used in the course of the study.
  Other Names: Viagra

SUMMARY:
Background: Intrapartum non-reassuring foetal status is a global challenge. It is a key contributor to operative deliveries. In low- and middle-income countries, it is a major cause of perinatal deaths, hypoxic ischemic encephalopathy, and cerebral palsy. Through its vasodilatory action and by improving uteroplacental perfusion, intrapartum sildenafil citrate could reduce the risk of intrapartum foetal compromise.

Aim: To determine the effect of intrapartum Sildenafil citrate on the prevention of non-reassuring foetal status among parturients delivering at term.

Specific Objectives: 1. To determine the frequency of non reassuring foetal heart rate (FHR) pattern among parturients delivering at term following administration of intrapartum Sildenafil citrate compared with placebo 2. To determine the rate of Caesarean delivery for non-reassuring FHR following the administration of intrapartum Sildenafil citrate compared with placebo. 3. To determine the rate of instrumental delivery for non-reassuring FHR following the administration of intrapartum Sildenafil citrate compared with placebo 4. To determine the effect of Sildenafil citrate on uteroplacental blood flow compared with placebo. 5. To determine if Sildenafil citrate is associated with an improved APGAR score at 5th minute compared with placebo.

Methodology: Study Design: Double blind randomised controlled trial. Women at term in early labour or undergoing scheduled induction of labour will be randomly allocated to receive 50 mg of sildenafil citrate or placebo orally once admitted in labour 6 hourly up to a maximum dose of 150 mg. Intrapartum foetal monitoring will be done by continuous cardiotocogragh, labour will be monitored with the aid of partograph following the departmental protocol for conduct of labour.

Planned Handling of Results: Obtained data will be analyzed using IBM (International Business Machines Corporation) SPSS (Statistical Product and Service Solutions) version 21, taking level of significance as p-value <0.05. Categorical variables will be expressed as percentages and presented using frequency tables and charts. The chi-square test will be used to test for association between categorical variables. Continuous variables will be presented as mean or median. Differences between continuous variables will be compared with the Student t test.

DETAILED DESCRIPTION:
Study Area The study will be carried out at LAUTECH Teaching Hospital (LTH), Ogbomoso. LTH Ogbomoso is located in Ogbomoso North Local Government area of Oyo state and most inhabitants are Yoruba speaking. It was officially commissioned in May, 2011. The study will be undertaken in the Obstetrics and Gynaecology Department of LTH Ogbomoso, the delivery rate in the department is about a hundred vaginal deliveries per month, average monthly antenatal clinic attendance of about two hundred and fifteen, an average annual caesarean section rate of 22.2% with foetal distress accounting for 14.0% of the cases was reported by Owonikoko et. al between 2011 and 2013.5

Study Design:

Double-blind, placebo-controlled, superiority randomised controlled trial.

Study Population Participants will be parturients with apparently uncomplicated, low-risk pregnancies, with appropriately grown foetuses, participants will be recruited at term (37-39+6 weeks of gestation). Women with both spontaneous and induced onset of labour will be considered eligible for inclusion. Those undergoing induction of labour will only be considered eligible if the indication for this was postdates pregnancy (before 42 weeks of gestation) or if induction had been planned for social reasons. Women undergoing induction as a result of foetal or maternal complications will not be included.

Recruitment of Participants:

All consented booked participants will be recruited at antenatal clinic at term (37+0 to 39+6 weeks). Participants shall be duly educated about the study procedure at the antenatal educational sessions. This information will be re-emphasised on arrival in labour ward.

Introduction of the study to the Participants:

The study procedure will be explained to the participants during antenatal education session as in appendix I (Information on the study procedure to participants) before the consent will be signed. Sufficient time will be afforded to potential participants to ensure they, and their support person (where applicable), can make an informed decision about their participation.

Data Collection After recruitment, selection of patients into each arm of the study will be through a computer generated sequence in a 1:1 ratio to receive either sildenafil citrate or placebo in variable blocks of up to six (Stata Statistical Software, Release 14; College Station, TX; StataCorp LP. StataCorp 2013) in a sealed opaque envelope. Each participant's study identification number will be recorded in the clinical notes and subsequently in their electronic health records.

The packaging of the trial drugs will be carried out under sterile hygienic condition in the hospital pharmacy department by two of the hospital pharmacists who will be dedicated to the study, they will prepare sequentially ordered packs labelled with individual study identification numbers containing identical tablets of sildenafil citrate or placebo, they will be the only one who know which number is assigned to sildenafil citrate or placebo. The same brand of sildenafil citrate (VIAGRA, manufactured by Fareva Amboise Zone Industrielle, 29 route des Industries, 37530 Poce Sur Cisse, France, under authority of Pfizer Inc, NewYork, NAFDAC Reg NO: 04 - 1509, Batch No: 477209; Exp date: 11 - 2024) will be used in the course of the study. The placebo will be a vitamin C of the same size, colour and shape with sildenafil (Viagra), this will be produced by TUYIL pharmaceutical company, Yidi road, Ilorin, Kwara state.

These will be stored in a locked drug cabinet in the birth suite. The midwife caring for each participant will then cross referenced the appropriate study pack with the study identification number recorded in the clinical notes and administered the trial tablet as specified in the protocol. Women, clinicians, and principal investigator will be unaware of allocation.

I (under the supervision of consultant radiologist) or a senior registrar in the department of radiology dedicated to the study will perform an ultrasound scan to measure indices of foetal and uteroplacental perfusion before and 2-4 hours after the initial dose of study medication.

An ultrasound scan will be performed to measure foetal biometry as well as Doppler resistance indices in the umbilical artery, umbilical vein, and middle cerebral artery. All ultrasound scans will be performed by me (principal investigator, under the supervision of consultant radiologist) or a senior registrar in the radiology department using a Voluson ultrasound machine with a 4- to 8-MHz curvilinear transabdominal transducer. To avoid caval compression, women will be positioned in a slightly left tilt supine position with the head of the bed elevated.

Clinical staff managing the labour will be blinded to the ultrasound results and retained responsibility for all decisions regarding intrapartum care. At LTH Ogbomoso, all decisions for caesarean delivery are made by the obstetrics team under the supervision of consultant Obstetrician.

Participants presenting for induction of labour, depending on the Modified Bishop's Score, induction of labour will be performed with balloon catheters or vaginal prostaglandin E1 analogue. In women with a favourable cervix, artificial rupture of membranes will be performed followed by an oxytocin infusion.

Women will receive the first dose of trial medication after transfer to the birth suite once diagnosed to be in labour with cervical dilatation < 8 cm. Sildenafil citrate will be given orally as a 50-mg dose 6 hourly to a maximum of 3 doses (150mg). Blood pressure will be monitored 15-30 minutes after each dose. Labour will be monitored with the aid of partograph, appropriate analgesic given in labour. Foetal heart rate monitoring will be performed in all cases by cardiotocograph or intermittent auscultation every fifteen minutes. Heart rate abnormalities will be classified using Royal College of Obstetricians and Gynaecologists (RCOG)/ National Institute for Clinical Excellence (NICE) categorisation of foetal heart rate feature.60 A Non-reassuring foetal heart rate pattern will be defined as one or more of the following features;60 Bradycardia, FHR <110 bpm Tachycardia, FHR > 160bpm Baseline variability < 5 bpm for 30 to 50 minutes OR More than 25 bpm for 15 to 25 minutes Absence of acceleration in 20 to 30 minutes tracing Early Deceleration Variable decelerations with no concerning characteristics* for 90 minutes or more OR Variable decelerations with any concerning characteristics* in up to 50% of contractions for 30 minutes or more OR Variable decelerations with any concerning characteristics* in over 50% of contractions for less than 30 minutes OR Late decelerations in over 50% of contractions for less than 30 minutes, with no maternal or foetal clinical risk factors such as vaginal bleeding or significant meconium

Subsidiary intrapartum and neonatal outcomes will include mode of birth (caesarean delivery, instrumental or spontaneous vaginal birth), indication for operative birth, length of labour (from time of active labour (cervical dilatation of > 4 cm to delivery of the infant), foetal heart rate abnormalities, meconium-stained liquor, postpartum haemorrhage (blood loss >500 mls), maternal intensive care unit admission, APGAR score at 5 minutes and, if admission to the special care baby unit (SCBU) occurred, length of stay, respiratory illness (transient tachypnoea of the newborn or pneumothorax), or neonatal encephalopathy.

Newborns will be screened for major Cardio-pulmonary disease and pulmonary hypertension by measuring oxygen saturation by pulse oximetry within 8 hours of birth.

Maternal symptoms potentially related to sildenafil citrate administration (nausea, vomiting, flushing, hypotension, blurred vision, visual loss, headache, dyspepsia, diarrhoea, and tremor) will be looked for and recorded.

All participants will be followed up within 48 hours of delivery. Medical records will be reviewed and intrapartum and neonatal outcome details recorded. The indication for operative delivery will be noted as recorded by the obstetric team.

In all cases, to ensure consistency of interpretation, intrapartum monitoring will be reviewed by two senior members of the obstetric team before a decision for intrapartum caesarean delivery for presumed foetal compromise will be performed.

Data Management The Proforma will be sorted out, entered into a computer and the obtained data will be analyzed using IBM (International Business Machines Corporation) SPSS (Statistical Product and Service Solutions) version 21. The method of data analysis will be as per-protocol i.e. data that will be included in the analysis will include only those participants who completed the treatment originally allocated to them as per protocol (data from participants who did not complete the treatment allocated to them or who did not comply with the protocol will not be included).

Categorical variables such as the socio-demographic status will be expressed as percentages and presented using frequency tables and charts. The chi-square test will be used to test for association between categorical variables on the contingency tables and statistical significance will be set at p values of less than 0.05.

Quantitative data e.g. gestational age will be presented as mean (standard deviation) or median (interquartile range). Differences between study groups will be compared with the Student t test and expressed as relative risk (RR), 95% confidence intervals (95% CIs). Ultrasound Doppler indices for MCA, UA, and cerebroplacental ratio will be converted to z scores using gestation-specific centiles,164 a p value of <0.05 will be deemed statistically significant.

Ethical Consideration The respondents will be informed that participation is voluntary and they will not suffer any consequence if they choose not to participate. All information gathered will be kept confidential. Participants will only be identified by hospital number without their name. Data obtained from the study will be stored in my personal passworded computer.

Ethical clearance will be obtained from the ethical committee of LTH Ogbomoso and permission will be obtained from the obstetrics and gynaecology head of department and Consultants staff to enrol their patients. All participants will receive written information about the study, it will be emphasized that the use of sildenafil citrate in labour is experimental and that it is not currently licensed for use for any obstetric indication. Sufficient time will be afforded to potential participants to ensure they, and their support person (where applicable), can make an informed decision about their participation and written informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Mother aged between 18- 49 years
2. Singleton pregnancy between 37+0 - 39+6 weeks gestation
3. Cephalic presentation
4. Foetus without any known structural, chromosomal or genetic abnormality
5. Planned vaginal delivery

Exclusion Criteria:

1. Women undergoing induction of labour as a result of foetal or maternal complications
2. Women in labour with Cervical dilatation > 8 cm,
3. Ruptured membranes with meconium stained liquor, or evidence of intrauterine infection.
4. Previous caesarean delivery
5. Foetus known to be small for gestational age, or suspected foetal growth restriction
6. Those with a contraindication to sildenafil citrate, such as hypersensitivity to sildenafil citrate, to an ingredient in its formulation, to nitrates or nitrites or to Riociguat.
7. Women with pre-existing heart disorders, stroke, hypotension or hypertension, pre-eclampsia, retinitis pigmentosa, kidney or liver abnormalities, sickle cell anaemia, gastrointestinal bleeding or any other bleeding disorder 40
8. Women taking any anti-hypertensive medication, alpha-adrenergic blocking agents, calcium channel blockers (verapamil), amyl nitrate, nicorandil, nitrates (including glyceryl trinitrate or isosorbide salts), sodium nitroprusside, bosentan, fosamprenavir and ritonavir combination, hepatic enzyme inhibitors CYP3A4 (including itraconazole, ketoconazole, ritonavir, cimetidine, erythromycin, saquinavir, darunavir), hepatic enzyme substrates (CYP3A4 and beta-adrenergic blocking agents), medications used to treat pulmonary arterial hypertension, and other phosphodiesterase type 5 inhibitors.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of non-reassuring foetal heart rate patterns | from admnistration of the drug till the delivery of the baby
  A Non-reassuring foetal heart rate pattern will be defined as one or more of the following features;60 Bradycardia, FHR <110 bpm Tachycardia, FHR > 160bpm Baseline variability < 5 bpm for 30 to 50 minutes OR More than 25 bpm for 15 to 25 minutes Absence of acceleration in 20 to 30 minutes tracing Early Deceleration Variable decelerations with no concerning characteristics* for 90 minutes or more OR Variable decelerations with any concerning characteristics* in up to 50% of contractions for 30 minutes or more OR Variable decelerations Late decelerations in over 50% of contractions for less than 30 minutes, with no maternal or foetal clinical risk factors such as vaginal bleeding or significant meconium
  * Regard the following as concerning characteristics of variable decelerations: lasting more than 60 seconds;

SECONDARY OUTCOMES:
Rate of emergency caesarean delivery for non-reassuring foetal status | at delivery
  rate of emergency caesarean section apart from non - reassuring foetal status
Rate of instrumental vaginal birth for non-reassuring foetal status | at delivery
  forceps delivery and vacuum delivery
Incidence of fresh meconium-stained liquor | from admnistration of the drug till the delivery of the baby
  greenish meconium liquor
Incidence of adverse neonatal outcomes ( APGAR score <7 at 5 minutes) | at delivery
  perinatal asphyxia
Rate of admission to the Special Care Baby Unit (SCBU) | at delivery
  any indications for admission to the special care baby unit at delivery
Incidence of neonatal encephalopathy (Sarnat stage 2 or 3) | at delivery
  hypoxic - ischaemic encephalopathy
Incidence of adverse maternal side effects | from admnistration of the drug till the delivery of the baby
  any side effects noticed in labour and delivery such as nausea, vomitting, headache

CONTACTS AND LOCATIONS:
Overall Officials: WAKEEL MURITALA, Principal Investigator — Ladoke Akintola University of Technology Teaching Hospital, Ogbomoso,Oyo State, Nigeria
Locations (1):
- Department of Obstetrics and Gynaecology, LAUTECH Teaching Hospital, Ogbomoso, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
proforma
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from 6 months